CLINICAL TRIAL: NCT05444231
Title: Breaking Through the Brain Fog: An Online RCT for Breast Cancer Survivors
Brief Title: Breaking Through the Brain Fog: An Online Research Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Dallas (Other)
Responsible Party: Principal Investigator, Sandra Chapman, PhD, Professor, The University of Texas at Dallas
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-434
Record Dates: First submitted 2022-06-29; First posted 2022-07-05 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer Female
Keywords: Cognitive Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Brain Training A (Experimental): This group will access one type of online brain-health oriented training.
  Interventions: Behavioral: Brain Training A
- Brain Training B (Active Comparator): This group will access a distinct type of online brain-health oriented training.
  Interventions: Behavioral: Brain Training B
- Brain Training C (Active Comparator): This group will access a distinct type of online brain-health oriented training.
  Interventions: Behavioral: Brain Training C

INTERVENTIONS:
Behavioral: Brain Training A — Interventions may include education, exercises, and/or strategies to support brain health
  Arms: Brain Training A
Behavioral: Brain Training B — Interventions may include education, exercises, and/or strategies to support brain health
  Arms: Brain Training B
Behavioral: Brain Training C — Interventions may include education, exercises, and/or strategies to support brain health
  Arms: Brain Training C

SUMMARY:
This study will investigate the benefits of distinct brain health trainings in breast cancer survivors (age 30-80) with cognitive concerns post-chemotherapy. This study can be completed from the comfort of participant's own home.

DETAILED DESCRIPTION:
Participants will complete online assessments at 3 timepoints over 6 months (Month 0, 3, 6). During the first 3 months of the study, participants will be randomized into one of three online training programs to support cognitive function; training will end after the first 3 months. The third online assessment (Month 6) will measure maintained gains since ending training. Participants will not be aware of the interventions assigned to other participants. Participants may be reimbursed for their time.

ELIGIBILITY:
Inclusion Criteria:

Female breast cancer survivors who...

* are between ages of 30-80
* were diagnosed with Stage I-III
* received chemotherapy
* completed chemotherapy at least 6 months ago but not more than 5 years
* endorse changes in thinking since end of chemotherapy treatment
* have working internet and a device
* consider themselves fluent in English

Exclusion criteria:

* Males
* A re-occurrence of breast cancer or a diagnosis of another
* An uncorrected hearing or vision issue that would hinder ability to read and/or listen to training material
* Participation in a cognitive training program in the last 12 months.
* A reported substance abuse problem
* Diagnosis of a neurodegenerative disease or psychotic disorder
* History of stroke, concussion, or brain injury since completing chemotherapy
* Inability to function independently due to Autism Spectrum Disorder diagnosis

Ages: 30 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2023-08-23 (Actual); Primary Completion 2025-03-09 (Actual); Study Completion 2025-03-09 (Actual)

PRIMARY OUTCOMES:
BrainHealth Index Score | Baseline, 3 month, 6 month
  The investigators will assess change on a holistic measure of cognitive, social, well-being, and daily life health on the BrainHealth Index across multiple timepoints. (Min value = 16, Max value = 1032) (Higher score = Better outcome)

SECONDARY OUTCOMES:
Functional Assessment of Cancer Therapy - Cognitive Function (FACT_Cog) | Baseline, 3 month, 6 month
  The investigators will assess change in self-reported cognitive deficits following an online training program. (Min value = 0, Max value = 148) (Higher score = better outcome)
Double Decision | Baseline, 3 month, 6 month
  The investigators will assess change scores on a visual processing speed task (Min value = 0, Max value = 100) (Higher score = Better performance)
Rapid Visual Information Processing | Baseline, 3 month, 6 month
  The investigators will assess change scores on measure of selective attention (Min value = 0, Max value = 100) (Higher score = Better performance)
Delayed matching to sample | Baseline, 3 month, 6 month
  The investigators will assess change scores on measure of visual memory (Min value = 0, Max value = 100) (Higher score = Better performance)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra B Chapman, PhD, Principal Investigator — Center for BrainHealth
Locations (1):
- The Center for BrainHealth at the University of Texas at Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chapman SB, Aslan S, Spence JS, Hart JJ Jr, Bartz EK, Didehbani N, Keebler MW, Gardner CM, Strain JF, DeFina LF, Lu H. Neural mechanisms of brain plasticity with complex cognitive training in healthy seniors. Cereb Cortex. 2015 Feb;25(2):396-405. doi: 10.1093/cercor/bht234. Epub 2013 Aug 28. PMID 23985135
- [Background] Chapman SB, Fratantoni JM, Robertson IH, D'Esposito M, Ling GSF, Zientz J, Vernon S, Venza E, Cook LG, Tate A, Spence JS. A Novel BrainHealth Index Prototype Improved by Telehealth-Delivered Training During COVID-19. Front Public Health. 2021 Mar 16;9:641754. doi: 10.3389/fpubh.2021.641754. eCollection 2021. PMID 33796498
- [Background] Chapman SB, Mudar RA. Enhancement of cognitive and neural functions through complex reasoning training: evidence from normal and clinical populations. Front Syst Neurosci. 2014 Apr 28;8:69. doi: 10.3389/fnsys.2014.00069. eCollection 2014. PMID 24808834
- [Background] Chapman SB, Aslan S, Spence JS, Keebler MW, DeFina LF, Didehbani N, Perez AM, Lu H, D'Esposito M. Distinct Brain and Behavioral Benefits from Cognitive vs. Physical Training: A Randomized Trial in Aging Adults. Front Hum Neurosci. 2016 Jul 18;10:338. doi: 10.3389/fnhum.2016.00338. eCollection 2016. PMID 27462210
- [Background] Chapman SB, Spence JS, Aslan S, Keebler MW. Enhancing Innovation and Underlying Neural Mechanisms Via Cognitive Training in Healthy Older Adults. Front Aging Neurosci. 2017 Oct 9;9:314. doi: 10.3389/fnagi.2017.00314. eCollection 2017. PMID 29062276
- [Background] Motes MA, Yezhuvath US, Aslan S, Spence JS, Rypma B, Chapman SB. Higher-order cognitive training effects on processing speed-related neural activity: a randomized trial. Neurobiol Aging. 2018 Feb;62:72-81. doi: 10.1016/j.neurobiolaging.2017.10.003. Epub 2017 Oct 12. PMID 29121545
- [Background] Han K, Davis RA, Chapman SB, Krawczyk DC. Strategy-based reasoning training modulates cortical thickness and resting-state functional connectivity in adults with chronic traumatic brain injury. Brain Behav. 2017 Apr 10;7(5):e00687. doi: 10.1002/brb3.687. eCollection 2017 May. PMID 28523229
- [Background] Vas A, Chapman S, Aslan S, Spence J, Keebler M, Rodriguez-Larrain G, Rodgers B, Jantz T, Martinez D, Rakic J, Krawczyk D. Reasoning training in veteran and civilian traumatic brain injury with persistent mild impairment. Neuropsychol Rehabil. 2016 Aug;26(4):502-31. doi: 10.1080/09602011.2015.1044013. Epub 2015 May 27. PMID 26018041
- [Background] Das N, Spence JS, Aslan S, Vanneste S, Mudar R, Rackley A, Quiceno M, Chapman SB. Cognitive Training and Transcranial Direct Current Stimulation in Mild Cognitive Impairment: A Randomized Pilot Trial. Front Neurosci. 2019 Apr 12;13:307. doi: 10.3389/fnins.2019.00307. eCollection 2019. PMID 31031581
- [Background] Han K, Martinez D, Chapman SB, Krawczyk DC. Neural correlates of reduced depressive symptoms following cognitive training for chronic traumatic brain injury. Hum Brain Mapp. 2018 Jul;39(7):2955-2971. doi: 10.1002/hbm.24052. Epub 2018 Mar 23. PMID 29573026
- [Background] Venza EE, Chapman SB, Aslan S, Zientz JE, Tyler DL, Spence JS. Enhancing Executive Function and Neural Health in Bipolar Disorder through Reasoning Training. Front Psychol. 2016 Nov 1;7:1676. doi: 10.3389/fpsyg.2016.01676. eCollection 2016. PMID 27847486